CLINICAL TRIAL: NCT06085001
Title: Lumella is a Point of Care Blood Test Used Together With Other Blood Tests to Assess the Risk of Preeclampsia in Pregnancy in 10 Minutes. Measurements of the Biomarker.
Brief Title: Use of Lumella-glycosylated Fibronectin for Diagnosis of Preeclampsia
Acronym: Lumella
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Croydon University Hospital (Other)
Responsible Party: Principal Investigator, Bini Ajay, Consultant Obstetrician and Gynaecologist, Croydon University Hospital
Other Study IDs: 329116
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Preeclampsia; Pregnancy Related; Hypertension
Keywords: Preeclampsia; PET
MeSH Terms: conditions — Pre-Eclampsia; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with preeclampsia: women with symptoms of preeclampsia from antenatal clinic or triage will be offered Lumella test along with traditional blood tests. If Lumella test is positive which will be compared with the traditional blood test results. Once 50 positive cases have been analysed the study results will be submitted to NICE.
  Interventions: Diagnostic Test: Lumella finger prick blood test

INTERVENTIONS:
Diagnostic Test: Lumella finger prick blood test — Finger prick blood test

SUMMARY:
women with symptoms of preeclampsia from antenatal clinic or triage will be offered Lumella test along with traditional blood tests. If Lumella test is positive which will be compared with the traditional blood test results. Once 50 positive cases have been analysed the study results will be submitted to NICE.

DETAILED DESCRIPTION:
Pre-eclampsia is a potentially serious condition that affects pregnant women. It is usually diagnosed during routine antenatal appointments. This is based on blood pressure measurements and results of urine protein tests that are recommended at each routine antenatal visit to screen for the condition. The Triage PlGF test and the Elecsys immunoassay sFlt-1/PlGF ratio is also recommended to help rule out the condition in women presenting with suspected pre-eclampsia between 20 weeks and 34 weeks of pregnancy plus 6 days. If diagnosed with pre-eclampsia, women are usually referred to a specialist in hospital for further tests and more frequent monitoring. Depending on the severity of the condition, some women may be monitored as outpatients while others may need admission to hospital for closer monitoring or to have the condition managed in a critical care setting.

The Lumella test is based on the novel biomarker GlyFn. The company states that compared with other currently used biomarkers (such as soluble fms-like tyrosine kinase-1 [sfIT-1] and placental growth factor [PlGF] or PlGF alone), GlyFn is etiological to pre-eclampsia and maintains a linear progression throughout pregnancy. The company also claims that the test offers improved sensitivity and specificity over standard care tests. This would lead to a reduction in false positives and false negatives. The Lumella test requires a finger prick blood sample (5 microlitres). Other pre-eclampsia tests currently used in the NHS need a phlebotomy blood sample, which can be difficult to collect in some people. The test can also be transported and stored at room temperature. Other tests for pre-eclampsia need to be refrigerated and brought to room temperature before the test can be done. The Lumella test may improve patient experience and allow a more rapid turnaround time for results. The company states that Lumella is currently the only test that can be done within 10 minutes at room temperature.

ELIGIBILITY:
Inclusion Criteria:

* If they can speak English
* Can give informed consent
* Has symptoms of Preeclampsia

Exclusion Criteria:

* Can't speak English
* Does not want to participate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant Women
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
can we use a bedside test -glycosylated fibronectin for the early diagnosis of pre-eclampsia | 6 months
  Does the test work?

SECONDARY OUTCOMES:
Is glycosylated fibronectin better than placental growth factor or traditional blood tests | 6 months
  Is the test better than PLGF/traditional blood tests

CONTACTS AND LOCATIONS:
Overall Officials: Bini Ajay, Principal Investigator — Croydon University Hospital
Locations (1):
- Croydon University Hospital, Croydon, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not sharing identifiable data

REFERENCES:
- See also: Huhn et al. BMC Pregnancy and Childbirth (2020) 20:128 https://doi.org/10.1186/s12884-020-2809-2 — http://doi.org/10.1186/s12884-020-2809-2
- See also: AM J Obstet Gynecol 2015;212:82.e1-9 Maternal Serum glycosylated fibronectin as a point-of-care biomarker for assessment of preeclampsia — https://doi.org/10.1016/j.ajog.2014.07.052